CLINICAL TRIAL: NCT03569683
Title: Efficacy of Low-level Laser Therapy, Hyaluronic Acid Gel and Herbal Gel as Adjunctive Tools in Gingivectomy Wound Healing-A Randomised Comparative Clinical and Histological Study
Brief Title: Comparison Between Laser, Synthetic Gel and Herbal Gel as Topical Agents After Gum Surgery
Acronym: CLSHGTAGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, Dr. Sana priyanka, Student, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMVIDS; 16201105032D (Other: Kaloji Narayana Rao University of Health Sciences.)
Record Dates: First submitted 2018-05-29; First posted 2018-06-26 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Gingival Overgrowth
MeSH Terms: conditions — Gingival Overgrowth | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: The patients will be equally divided into three groups. (Groups A,B&C) All the cases will be prepared preoperatively with scaling and root planing, oral hygeine instructions, occlusal equilibration and dietary evaluation. External bevel gingivectomy will be performed wherein the inflamed gingiva will be excised and shaped.
  Group A- The Surgical site will be treated with diode laser following gingivectomy procedure, immediately and on the 1st,3rd and 7th day after surgery.
  Group B- Hyaluronic acid will be applied topically to the surgical site immediately after gingivectomy, tin foil would be placed and periodontal dressing given, and on the 1st,3rd and 7th day postoperatively.
  Group C- Herbal gel will be applied topically and tin foil placed over which a periodontal dressing would be given immediately after the surgery and on the 1st,3rd and 7th day postoperatively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional Single arm (Experimental): Group A- Diode laser biostimulation on surgical site immediately after external bevel gingivectomy and on 1st,3rd, and 7th day after surgery.
  Group B- Hyaluronic acid (Gengigel) topical application on surgical site immediately after external bevel gingivectomy and on 1st,3rd, and 7th day after surgery.
  Group C- Herbal gel (Hiora SG) topical application on surgical site immediately after external bevel gingivectomy and on 1st,3rd, and 7th day after surgery.
  Interventions: Procedure: External bevel gingivectomy; Device: Diode laser Biostimulation; Other: Hyaluronic acid (Gengigel) topical application.; Other: Herbal gel (Hiora SG) topical application

INTERVENTIONS:
Procedure: External bevel gingivectomy — External bevel gingivectomy will be performed on 30 patients wherein the suprabony pockets will be eliminated with the help of a Bard parker blade no 15. The incision would be given 1mm apical to the pockets which would be marked by a Crane and Kaplan pocket marker, then the incision would be given and the tissue would be removed with the help of kirkland and orbans knives and the gingiva would be shaped. After the surgical procedure the patients would be treated either with the Diode laser(Group A), Hyaluronic acid gel (Group B), or Herbal gel(Group C).
  Other Names: Conventional Gingivectomy
Device: Diode laser Biostimulation — After gingivectomy, laser irradiation will be done using bio-stimulation tip in the anterior sextants of the mouth. (Group A)
Other: Hyaluronic acid (Gengigel) topical application. — After gingivectomy, Hyaluronic acid gel(Gengigel) will be applied topically. Then it will be covered with a tin foil and periodontal dressing would be given. (Group B)
Other: Herbal gel (Hiora SG) topical application — After gingivectomy, Herbal gel(Hiora SG) will be applied topically. Then it will be covered with a tin foil and periodontal dressing would be given. (Group C)

SUMMARY:
This study would be conducted to assess the effectiveness of low-level laser therapy, hyaluronic acid gel and herbal gel as adjunctive aids in the healing of gingivectomy wounds. As the gingivectomy wound heals by secondary intention, this study aims to compare the healing potential of low-level laser therapy, hyaluronic acid gel and herbal gel when applied topically at baseline, 1st day,3rd day and 7th day after gingivectomy procedure.

DETAILED DESCRIPTION:
Low-level laser therapy applied to soft tissues stimulates specific metabolic processes in healing wounds. Major changes observed in wounds treated with low-level laser therapy(LLLT) include increased healthy granulation tissue formation with early epithelization, increased fibroblast proliferation and matrix synthesis.

Hyaluronic acid is a polysaccharide gel and it has many properties that make it a potentially ideal molecule for assisting in wound healing by inducing early granulation tissue formation, inhibiting inflammation, providing epithelial turnover and also aiding in connective tissue angiogenesis.

Hiora gel is a herbal astringent gel which helps in wound healing, reduces inflammation and also alleviates pain.

ELIGIBILITY:
Inclusion Criteria: Gingival enlargement index greater than or equal to 2mm

Exclusion Criteria: Infrabony Pockets Diabetic patients Smokers.

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Histological Assessment | Immediately Postoperatively and 6 weeks after gingivectomy.
  Change in gingival tissue healing will be assessed.0.5 mm of tissue will be taken from the interdental papilla distal to the canine and will be processed for examination using hematoxiline and eosin and picrosirus staining.

SECONDARY OUTCOMES:
Clinical Parameters | 6 weeks after Gingivectomy procedure
  Gingival tissue healing will be assessed on a 10 point visual analogue scale.Score in each tooth will be taken including one full interdental papilla
  Visual Analogue Scale: will be used to quantify pain levels and patient's discomfort. The VAS consists of a horizontal line of 10 cm (100 mm) with two end-points representing 'no pain' and 'worst pain imaginable'. Patients will be asked to rate their pain by placing a mark on the line corresponding to their current level of pain. The distance along the line from the 'no pain' marker is then measured with a ruler giving a pain score out of 10.
  0: No pain 1-3: Slight pain 3.1-6: Moderate pain 6.1-10: Severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Priyanka Reddy, (MDS), Principal Investigator — PG Student
Locations (1):
- Panineeya Mahavidyalaya Institute of Dental Sciences and Research Centre, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amorim JC, de Sousa GR, de Barros Silveira L, Prates RA, Pinotti M, Ribeiro MS. Clinical study of the gingiva healing after gingivectomy and low-level laser therapy. Photomed Laser Surg. 2006 Oct;24(5):588-94. doi: 10.1089/pho.2006.24.588. PMID 17069488
- [Background] Martu S, Amalinei C, Tatarciuc M, Rotaru M, Potarnichie O, Liliac L, Caruntu ID. Healing process and laser therapy in the superficial periodontium: a histological study. Rom J Morphol Embryol. 2012;53(1):111-6. PMID 22395509